CLINICAL TRIAL: NCT03021759
Title: Pragmatic, Randomized Evaluation of Statin Active Choice to Reach Improved Outcomes Based on Evidence
Acronym: PRESCRIBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 826125
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- Active choice (Experimental): Physicians will be asked to review a list of their patients eligible for statin therapy who are not yet prescribed a statin and make an active choice whether or not to prescribe a statin.
  Interventions: Behavioral: Active choice
- Active choice with social comparison feedback (Experimental): Physicians will be asked to review a list of their patients eligible for statin therapy who are not yet prescribed a statin and make an active choice whether or not to prescribe a statin. Physicians will receive social comparison feedback informing them of how their performance compares to their peers
  Interventions: Behavioral: Active choice; Behavioral: Social comparison feedback

INTERVENTIONS:
Behavioral: Active choice — Statin options are framed to physicians as an active choice to prescribe or not prescribe a statin
  Arms: Active choice; Active choice with social comparison feedback
Behavioral: Social comparison feedback — Statin prescribing rates are communicated to physicians and along with how their performance compares to their peers
  Arms: Active choice with social comparison feedback

SUMMARY:
In this study, the investigators will conduct a pragmatic, cluster-randomized, controlled trial to evaluate an active choice intervention with and without social comparison feedback to increase physician statin prescribing rates for eligible patients.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in the United States. Strong evidence indicates that statin medications can reduce the risk of CVD and for those with CVD statins have been shown to reduce mortality. Despite this evidence, statins are under-prescribed. In this study, the investigators will test the effectiveness of nudges targeted to physicians using active choice and social comparisons feedback to increasing the rate at which statin medications are prescribed to patients eligible based on national practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a primary care physician at University of Pennsylvania Health System
* Patient meets 2013 AHA/ACC guidelines for statin therapy but no record of a statin prescription in the electronic health record

Exclusion Criteria:

* Patient has an allergy or adverse reaction to statins documented in the electronic health record
* Patient has glomerular filtration rate less than 30 mL/min
* Physicians (and their respective patients) will be excluded if they have less than 10 patients among their entire panel that are eligible for a statin

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4774 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Patel MS, Kurtzman GW, Kannan S, Small DS, Morris A, Honeywell S Jr, Leri D, Rareshide CAL, Day SC, Mahoney KB, Volpp KG, Asch DA. Effect of an Automated Patient Dashboard Using Active Choice and Peer Comparison Performance Feedback to Physicians on Statin Prescribing: The PRESCRIBE Cluster Randomized Clinical Trial. JAMA Netw Open. 2018 Jul 6;1(3):e180818. doi: 10.1001/jamanetworkopen.2018.0818. PMID 30646039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No informed consent was obtained from the participants in this study.
Period: Overall Study
Arm/Group | Control | Active Choice | Active Choice With Social Comparison Feedback
Started | 1566 | 1743 | 1465
Completed | 1566 (32 primary care physicians were randomized to this arm and analyzed.) | 1743 (32 primary care physicians were randomized to this arm and analyzed.) | 1465 (32 primary care physicians were randomized to this arm and analyzed.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Active Choice | Active Choice With Social Comparison Feedback | Total
Number analyzed (Participants) | 1566 | 1743 | 1465 | 4774
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (8.5) | 62.4 (8.2) | 62.5 (8.2) | 62.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 738 | 710 | 701 | 2149
  Male | 828 | 1033 | 764 | 2625
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 1004 | 1110 | 926 | 3040
  Black non-Hispanic | 420 | 479 | 419 | 1318
  Other | 142 | 154 | 120 | 416
Annual Household Income [Count of Participants; unit: Participants]
  <50,000 US$ | 435 | 563 | 406 | 1404
  50,000 - 100,000 US$ | 784 | 960 | 733 | 2477
  >100,000 US$ | 341 | 206 | 312 | 859
  Missing | 6 | 14 | 14 | 34

OUTCOME MEASURES:

1. Primary Outcome: Statin Prescribing Rate
Description: Percentage of patients eligible for a statin that have been prescribed a statin
Time Frame: Two Months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Active Choice | Active Choice With Social Comparison Feedback
Number analyzed (Participants) | 1566 | 1743 | 1465
Participants | 40 | 116 | 117

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Control | Active Choice | Active Choice With Social Comparison Feedback
All-Cause Mortality (participants affected / at risk) | 0/1566 | 0/1743 | 0/1465
Serious Adverse Events (participants affected / at risk) | 0/1566 | 0/1743 | 0/1465
Other Adverse Events (participants affected / at risk) | 0/1566 | 0/1743 | 0/1465

LIMITATIONS AND CAVEATS:
Physicians and patients were from a single health care system and we did not have data on prescription fill rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03021759/Prot_SAP_000.pdf